CLINICAL TRIAL: NCT02813746
Title: Maternal Transcriptomic Regulation of the Preimplantation Embryo
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Igenomix (Industry)
Responsible Party: Principal Investigator, Carlos Simon, Scientific Director IGENOMIX; Gynaecologist IVI Valencia, Igenomix
Other Study IDs: 1603-IGX-018-CS
Record Dates: First submitted 2016-06-22; First posted 2016-06-27 (Estimated); Last update posted 2016-06-28 (Estimated); Status verified 2016-06

CONDITIONS: Fetal Origin of Adult Diseases
Keywords: Obesity; Tobacco; Epigenetic; Transcriptomic; microRNAs; miRNAs
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA will be analyzed in the endometrial fluid. These samples will be completely exhausted during the analysis.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Obese non smoker vs Normoweight non smoker: Endometrial fluid (EF) will be obtained from non-smokers normo-weight and obese patients in the receptive state. Samples will be collected 7 days after Luteinizing Hormone (LH) peak. They will be classified following the guidelines of the obesity classification system by the World Human Organization (WHO). Patients will be subjected to a fitness program during a year with the aim to achieve a weight reduction to normal values (19-24.9 kg/m2). The modifications in the miRNAs expression will be studied. After the weight loss, new EF will be collected from these patients.
  Interventions: Dietary Supplement: Fitness program; Procedure: Endometrial fluid collection
- Normoweight smoker vs Normoweight non-smoker: EF will be obtained from non-smokers and smokers normo-weight in the receptive state. Samples will be collected 7 days after Luteinizing Hormone (LH) peak. Smokers patients will be urge to give up smoking during at least one year. After this time, new samples will be collected to determine if the non-exposition to this contaminant could exert any effect in the miRNAs signature. A regular control will be done in this group of patients to ensure that they have not been exposed to tobacco in 12 months. Professional support will be given in the same centre of the study to help the patient to accomplish its objective.
  Interventions: Behavioral: Stop smoking; Procedure: Endometrial fluid collection

INTERVENTIONS:
Dietary Supplement: Fitness program
  Groups: Obese non smoker vs Normoweight non smoker
Behavioral: Stop smoking
  Groups: Normoweight smoker vs Normoweight non-smoker
Procedure: Endometrial fluid collection

SUMMARY:
The aim of this study is to understand the epigenetic and transcriptomic mechanisms that regulate the fetal origin of adult diseases (FOAD), either for the presence of metabolic disorders in the future mothers, such as obesity or for the exposure to certain contaminants such as tobacco.

To do that, the miRNAs profiles secreted to the endometrial fluid in obese women vs normoweight women during the window of implantation will be identified. Likewise, it will be studied how that miRNA signature is normalized once a substantial loss of weight is produced by the patients involved in the studied. In parallel, a comparison of the miRNA expression profiles secreted in the endometrial fluid in smoker women vs nonsmoker women will be performed. As in the previous case, it will be studied if after the exposure to these contaminant, the normalization of the miRNA expression signature occurs. Finally, an in silico analysis will be carried out in order to define the target genes and the metabolic pathways affected by the miRNAs profile secreted in both pathological conditions

DETAILED DESCRIPTION:
The developmental origins of adult disease are now recognized to be related to intrauterine conditions during embryonic and fetal life. Pregnancy begins with embryo implantation and its impact in adult life remains unknown. It has been demonstrated that human endometrial epithelium secretes specific microRNAs (miRNAs) during the time frame when the embryo enters the uterine cavity and initiates its adhesion to the uterine wall. Maternal miRNAs are secreted to the endometrial fluid, transported through exosomes or bound to proteins and consequently uptaken by the preimplantation embryo, before implantation occurs. As a consequence they suffer transcriptomic modifications that induce profound molecular and functional changes. The data already published demonstrate a novel paradigm: the transcriptomic maternal endometrial regulation of the pre-implantation embryo in health.

Here, this novel maternal endometrium-based mechanism will be applied in order to understand and prevent the developmental origin of adult diseases induced during embryonic implantation either by metabolic disorders of future mothers who have developed obesity or by the exposure to certain contaminants such as tobacco. In this project, the expression profiles of secreted miRNAs will be identified in the endometrial fluid in obese women compared to normo-weight women. Also, it will be studied how this "obese" endometrial miRNA pattern is reversed after weight-loss. In parallel, murine models of obesity will be used to proof this concept. In addition, the expression profiles of secreted endometrial miRNAs will be identified in smokers versus future non-smokers mothers. As in the previous case, the reversion of this signature will be analysed after stopping the exposure to this contaminant.

Then, "in silico" analysis will be done to select putative genes and functional pathways targeted by the signature of secreted endometrial miRNAs in the human and murine models in both pathological conditions. The determination of the transcriptomic and/or epigenome modifications induced by "obese" or/and "smoker" endometrial miRNAs in preimplantation mouse embryos is expected. As preliminary results, to support this project our accepted model of transcriptomic maternal endometrial regulation of the pre-implantation embryo in health, and the identification of a differential pattern of secreted miRNAs in the endometrial fluid of obese women compared to normo-weight counterparts is presented. In consequence, the application of this novel endometrium-based mechanism to the understanding and prevention of the origin of adult diseases related to obesity and/or tobacco exposure is proposed.

ELIGIBILITY:
Inclusion Criteria:

* Women with age comprised between 18 and 45 years
* Normal uterus (evaluated trough ultrasound 2D/3D and/or hysteroscopy)
* Presence of at least one ovary
* Body mass index:
* Normoweight: 18.0-24.9 kg/m2 and non smokers
* Obese ≥30.0 kg/m2 and non smokers
* Smokers: Normoweight and smoke at least 10 cigarettes per day

Exclusion Criteria:

* Overweight=25.0-29.9 kg/m2
* Patients with Intrauterine device in the last 3 months
* Patients who had had hormonal contraceptives in the 2 previous months.
* Adnexal or uterine pathologies
* Polycystic ovary
* Existence of serious or uncontrolled bacterial, fungal or viral infections that could interfere with the involvement of the patient in the study or in the evaluation of the study results.
* Any disease or medical condition that could be unstable or could endanger the security of the patient and her compliance in the study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Endometrial fluids from non-smoker obese and normoweight samples will be analysed in the window of implantation. In turn, endometrial fluids from normoweight smoker and non-smoker patients will be analysed in the window of implantation.
  These participants will be recruited in just one centre: IVI Valencia. Their recruitment will be done through a routine consultation carried out by the research team from the centre, as well as through the revision and daily evaluation of the medical reports and subsequent contact with those patients who could accomplish with the criteria selection and desire to be involved in the study.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-04 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Understanding of the epigenetic and transcriptomic mechanisms that regulate the FOAD | 40 months
  The main objective of the present project is focused on understanding the epigenetic and transcriptomic mechanisms that regulate the fetal origin of adult diseases (FOAD) either by the presence of metabolic disorders in mothers such as obesity, or by the exposure to certain pollutants such as tobacco

SECONDARY OUTCOMES:
Analysis of the miRNA expression pattern in the endometrial fluid (EF) in obese patients Analysis of the miRNA expression profile in the endometrial fluid | 13 months
  miRNA expression profile will be analysed in obese women , in comparison to normoweight women during the window of implantation. In turn, the normalization of this particular transcriptomic signature will be studied after the existence of a substantial loss of weight by the patients involved in the study.
Analysis of the miRNA expression pattern in the endometrial fluid (EF) in smoker patients | 13 months
  A comparison between the miRNA expression profiles in smoker women vs. non-smoker will be done in the endometrial fluid (EF) during the window of implantation. As in the previous case, it will be studied if that particular pattern is normalized after giving up smoking.
Functional analysis | 13 months
  The target genes and the metabolic routes affected by the miRNA profile secreted in both pathological conditions will be defined.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Simón, MD PhD, Principal Investigator — Igenomix
Locations (1):
- IVI Valencia, Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No